CLINICAL TRIAL: NCT06988982
Title: Lipid Emulsion for Reversal of Spinal Anesthesia in Ambulatory Surgery: A Randomized Controlled Trial
Brief Title: Lipid Emulsion for Reversal of Spinal Anesthesia in Ambulatory Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Associate professor of anesthesia, intensive care, and pain management, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1270/13-5-2025
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Spinal Anaesthesia; Spinal Anesthesia Evaluation; Ambulatory Surgery
Keywords: lipid emulsion; spinal anesthesia; ambulatory surgery
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ILE (Intravenous lipid emulsion group) (Experimental): patients will receive 1.5 ml/kg bolus of intravenous lipid emulsion 20 % followed by 0.25 ml/kg/hour infusion over 30 minutes at the end of surgery
  Interventions: Drug: Intravenous Lipid Emulsion 20%
- Group C (control group) (Placebo Comparator): patients will received equal volume of normal saline at the end of surgery
  Interventions: Drug: Control (placebo) group

INTERVENTIONS:
Drug: Intravenous Lipid Emulsion 20% — patients will receive 1.5 ml/kg bolus of intravenous lipid emulsion 20 % followed by 0.25 ml/kg/hr infusion over 30 minutes at the end of surgery
  Arms: Group ILE (Intravenous lipid emulsion group)
Drug: Control (placebo) group — patients will receive equal volume of normal saline at the end of surgery
  Arms: Group C (control group)

SUMMARY:
Ambulatory surgery places high demands on anesthetic technique. rapid onset and offset of anesthesia, rapid recovery of protective reflexes, mobility and micturition, are required. Since the inception of ambulatory surgery, the favored anesthetic technique has been general anesthesia with short-acting drugs. Concerns about the time to perform spinal anesthesia and the risks of prolonged motor block and urinary retention have limited its use.

Alpha-blockers, lavage fluids for epidural space, insulin, and intravenous lipid emulsions, are still being discussed to shorten and reverse adverse effect of different LAs used for spinal anaesthesia, hence we will evaluate the effectiveness of intravenous lipid emulsion for reversing the neural blockade of spinal anaesthesia in patients undergoing ambulatory surgery.

DETAILED DESCRIPTION:
An increasing number of ambulatory surgical patients is challenging the currently used anaesthesia methods, reliable surgical anaesthesia should be quick, with rapid recovery and minimal side effects. Spinal anaesthesia (SA) is an easy and reliable technique that has grown in popularity for inpatient surgery, but its use in ambulatory surgery has been limited due to several factors including the prolonged neurological block with long-acting local anaesthetics (LA), delayed ambulation, risk of urinary retention and pain after block regression therefore delaying patient discharge. On the other hand, general anaesthesia with short-acting drugs grants rapid recovery enabling the early discharge. While recovery after spinal anaesthesia has been recently improved by lowering the dose of the commonly used long-acting local anaesthetics such as bupivacaine, discharge times are still prolonged compared to general anaesthesia.

Intravenous lipid emulsions (ILEs) were originally developed as a part of parenteral nutrition for critically ill patients, dating back to the 1960s. Over the last ten years, there has been rising interest in ILEs in clinical toxicology beyond its established role in the treatment of acute intoxication with local anaesthetics (LAST). The use of ILEs for the treatment of lipophilic drug toxicity is increasing nowadays with several studies reported alleviation of intractable cardiovascular collapse induced by toxic doses of these non-local anaesthetic drugs including calcium channel blockers (verapamil), tricyclic antidepressants (amitriptyline) and beta-blockers. In addition, Complications following intrathecal administration of bupivacaine have been reported to be successfully managed with intravenous administration of lipid emulsion.

While the precise mechanism by which ILEs exerts its effect remains unknown, the leading theory is that the ILEs intravascular action entails creating a concentration gradient which favours LA redistribution to the extracellular space. Lipid vesicles then encapsulate LA creating lipid sinks and the formation of this "trap" removes the toxins from the various tissues and organs, reducing their bioavailability and the sequestration mechanism where LA is rapidly redistributed by "lipid shuttles" to sites of metabolism (liver), storage (adipose tissue) or elimination (kidney). Alternative theories include reduced binding of local anaesthetics to sodium transport channels, direct promotion of sodium channel function recovery, and replenishing ATP stores from increased uptake of fatty acids by mitochondria.

Considering the few published reports supporting the effectiveness of ILEs in reversing the primary nervous system effects of regional anaesthesia such as total or high spinal anaesthesia, prolonged neural blockade, and reverse phrenic nerve palsy secondary to a brachial plexus block with the well-known favourable safety profile of ILEs. We hypothesized that ILEs could be an attractive effective option to reverse the sensory and motor actions of intrathecal bupivacaine thus accelerating the neurological recovery after spinal anaesthesia which could avert the delayed hospital discharge and facilitate the use of SA for ambulatory surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Cooperative patient
* Age 21-70 years old.
* BMI ≤ 35 kg/m2
* ASA I - II.
* Elective ambulatory surgery under spinal anesthesia (general surgery, urology, gynecology, orthopedic surgery).

Exclusion Criteria:

* History of allergy to the LA agents used in this study,
* Skin lesion at needle insertion site,
* Those with bleeding disorders, sepsis, liver disease and psychiatric disorders
* History of cognitive dysfunction or mental illness

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Time for complete sensory and motor regression (min) | 6 hours after surgery
  Time for complete sensory regression (min) (primary outcome) to be calculated from the time of ILEs administration (T0) until full sensation at S1 dermatomal level achieved Time for complete motor regression (min) (primary outcome) to be calculated from time of ILEs administration (T0) until Bromage score will be zero.

SECONDARY OUTCOMES:
Time for two segment sensory regression (min) | 6 hours after surgery
  the time for regression by two dermatomes compared with the dermatomal level assessed at finishing ILEs infusion (T0)
Time to walk (min) without or with minimal assistance | 6 hours after surgery
  the time from the ILE administration time (T0) till the patients first stand and walk.
Time to Void (min) | 6 hours after surgery
  the time from the ILE administration time (T0) till the patients first urinate.
Time to be home-ready (min) | 6 hours after surgery
  the time from the ILE administration time (T0) till the patients are ready for home discharge as defined by the modified post anaesthesia discharge scoring system.
Time to actual hospital discharge (min) | 24 hours after surgery
  the period from the end of the surgery till the patients actually leaves the hospital.
Heart rate (HR), and arterial blood pressure (MAP) | 6 hours after surgery
  Heart rate (HR), and arterial blood pressure (MAP), will be recorded immediately before and after the ILEs administration, at PACU admission and then every 15 min till the PACU discharge.
Numerical rating scale (NRS) | 24 hours after surgery
  Numerical rating scale (NRS) will be postoperatively assessed and recorded at PACU admission, PACU discharge to phase II recovery, in phase II recovery room, before actual hospital discharge and at 24 h.
Time to first rescue analgesia (min) | 24 hours after surgery
  the time between ILE administration (T0) to the time patients make their first request for pain relief and NRS ≥ 3.
Total dose of rescue analgesia (diclofenac sodium) | 24 hours after surgery
  Total dose of rescue analgesia (diclofenac sodium), that will be consumed in the first 24 hours postoperatively.
Postoperative Complications. | 2 weeks after surgery
  Postoperative complications will be evaluated including nausea and vomiting, the use of antiemetics, inability to void within 4h after surgery, post-dural puncture headache, transient neurological symptoms (TNS) and lipid emulsions related adverse effects such as hypotension, bradycardia, fever, dyspnea, allergic reaction, increased risk of infection, and fat overload syndrome.
  The day after surgery and for one week, all patients will be contacted by telephone and asked about pain and analgesic use, low back pain, headache and transient neurological symptoms. One and two weeks after surgery, patients will be evaluated by the surgical team and the existence of any complications will be recorded.
Patient satisfaction | 2 weeks after surgery
  Patient satisfaction using a 3-point Likert scale (3=satisfied, 2= neutral, 1=dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M. S. Mowafy, MD, Principal Investigator — Anaesthesia, Intensive Care, and Pain Management Department. Faculty of Medicine, Zagazig University,; Shereen E. Abd Ellatif, MD, Study Director — Anaesthesia, Intensive Care, and Pain Management Department. Faculty of Medicine, Zagazig University
Locations (1):
- Zagazig University Hospitals, Zagazig, Al Sharqia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available 6 months after publication
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Palumbo P, Tellan G, Perotti B, Pacile MA, Vietri F, Illuminati G. Modified PADSS (Post Anaesthetic Discharge Scoring System) for monitoring outpatients discharge. Ann Ital Chir. 2013 Nov-Dec;84(6):661-5. PMID 23165318
- [Background] Bromage PR. A comparison of the hydrochloride and carbon dioxide salts of lidocaine and prilocaine in epidural analgesia. Acta Anaesthesiol Scand Suppl. 1965;16:55-69. doi: 10.1111/j.1399-6576.1965.tb00523.x. No abstract available. PMID 5322004
- [Background] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Background] 14. Kumar KS, Talawar P, Gupta B, et al. OP020 Efficacy of 20% intravenous lipid emulsion as a reversal agent of spinal anaesthesia: a double blinded randomized controlled trial. Regional Anesthesia & Pain Medicine 2023;48:A12.
- [Background] Tampakis K, Vogiatzakis N, Kontogiannis C, Spartalis M, Ntalianis A, Spartalis E, Siafaka I, Iacovidou N, Chalkias A, Xanthos T. Intravenous lipid emulsion as an antidote in clinical toxicology: a systematic review. Eur Rev Med Pharmacol Sci. 2020 Jun;24(12):7138-7148. doi: 10.26355/eurrev_202006_21708. PMID 32633409
- [Background] Cave G, Harvey M, Graudins A. Intravenous lipid emulsion as antidote: a summary of published human experience. Emerg Med Australas. 2011 Apr;23(2):123-41. doi: 10.1111/j.1742-6723.2011.01398.x. Epub 2011 Apr 7. PMID 21489160
- [Background] 11. Hadbi M, Benalakma D, Berbiche R, et al. Effect of lipid infusion on the reversal of atypically prolonged duration and high spinal anesthesia. About two cases. J Clin Res Anesthesiol. 2021; 4: 1-4.
- [Background] 10. Hadbi M, Benalakma D, Berbiche R, et al. Abnormal Prolonged Duration of Spinal Anesthesia in Patient with Multiple Sclerosis. J Anesth Clin Res. 2021; 12: 984.
- [Background] 9. Joseph Eldor, Pham V, Tran TP, et al. Local Anesthesia Reversal LAR of Total Spinal Anesthesia TSA by Lipofundin Lipid Emulsion. Jor Health Sci Development. 2018; 1: 67-72.
- [Background] 8. Seglenieks R, Chowdhury A. Use of Lipid Emulsion to Reverse the Effects of Regional Anesthesia: A Novel Indication. Translational Perioperative and Pain Medicine. 2023; 10 (1):512-514. DOI 10.31480/2330-4871/171.
- [Background] Hoshino R, Kamiya Y, Fujii Y, Tsubokawa T. Lipid emulsion injection-induced reversal of cardiac toxicity and acceleration of emergence from general anesthesia after scalp infiltration of a local anesthetic: a case report. JA Clin Rep. 2017;3(1):9. doi: 10.1186/s40981-017-0077-6. Epub 2017 Feb 10. PMID 29492448
- [Background] Muller SH, Diaz JH, Kaye AD. Clinical applications of intravenous lipid emulsion therapy. J Anesth. 2015 Dec;29(6):920-6. doi: 10.1007/s00540-015-2036-6. Epub 2015 Jun 7. PMID 26049929
- [Background] Picard J, Meek T. Lipid emulsion for intoxication by local anaesthetic: sunken sink? Anaesthesia. 2016 Aug;71(8):879-82. doi: 10.1111/anae.13395. Epub 2016 Feb 8. No abstract available. PMID 26854285
- [Background] Afolayan JM, Olajumoke TO, Olaogun J, Kadiri I. Reversal of spinal anaesthesia and prevention of post operative complications using intralipid emulsion. J Clin Images Med Case Rep. 2024; 5(2): 2880.
- [Background] Waring WS. Intravenous lipid administration for drug-induced toxicity: a critical review of the existing data. Expert Rev Clin Pharmacol. 2012 Jul;5(4):437-44. doi: 10.1586/ecp.12.27. PMID 22943123
- [Background] Ok SH, Hong JM, Lee SH, Sohn JT. Lipid Emulsion for Treating Local Anesthetic Systemic Toxicity. Int J Med Sci. 2018 May 14;15(7):713-722. doi: 10.7150/ijms.22643. eCollection 2018. PMID 29910676
- [Background] Rattenberry W, Hertling A, Erskine R. Spinal anaesthesia for ambulatory surgery. BJA Educ. 2019 Oct;19(10):321-328. doi: 10.1016/j.bjae.2019.06.001. Epub 2019 Aug 13. No abstract available. PMID 33456853